CLINICAL TRIAL: NCT05690061
Title: Effects of Different Sources of Beef and Plant-based Meat Alternatives on Postprandial Inflammatory and Metabolic Profiles of Consumers
Brief Title: Beef and Plant Burger Metabolomics Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: Duke University (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephanvanvliet, Principal Investigator, Utah State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 12499
Record Dates: First submitted 2022-12-19; First posted 2023-01-19 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Response
Keywords: Metabolomics; Human Nutrition; Meat; Plant-based Meat Alternative

STUDY DESIGN:
Intervention Model Description: Randomized cross-over design with 250 g of cooked meat (grain-fed hamburger, grass-fed hamburger, Impossible Burger) ingested and blood draws, urine, and questionnaires collected on separate visits.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which type of burger they consume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1: Grain-Fed, Grass-Fed, Impossible (Active Comparator): On the first visit, a grain-fed beef burger (250 grams) will be consumed.
  On the second visit, a grass-fed beef burger (250 grams) will be consumed.
  On the third visit, an Impossible BurgerTM (250 grams) will be consumed.
  Interventions: Dietary Supplement: Grain-Fed Beef Hamburger; Dietary Supplement: Grass-Fed Beef Hamburger; Dietary Supplement: Impossible BurgerTM
- Sequence 2: Grass-Fed, Grain-Fed, Impossible (Active Comparator): On the first visit, a grass-fed beef burger (250 grams) will be consumed.
  On the second visit, a grain-fed beef burger (250 grams) will be consumed.
  On the third visit, an Impossible BurgerTM (250 grams) will be consumed.
  Interventions: Dietary Supplement: Grain-Fed Beef Hamburger; Dietary Supplement: Grass-Fed Beef Hamburger; Dietary Supplement: Impossible BurgerTM
- Sequence 3: Impossible, Grass-Fed, Grain-Fed (Active Comparator): On the first visit, an Impossible BurgerTM (250 grams) will be consumed.
  On the second visit, a grass-fed beef burger (250 grams) will be consumed.
  On the third visit, a grain-fed beef burger (250 grams) will be consumed.
  Interventions: Dietary Supplement: Grain-Fed Beef Hamburger; Dietary Supplement: Grass-Fed Beef Hamburger; Dietary Supplement: Impossible BurgerTM
- Sequence 4: Impossible, Grain-Fed, Grass-Fed (Active Comparator): On the first visit, an Impossible BurgerTM (250 grams) will be consumed.
  On the second visit, a grain-fed beef burger (250 grams) will be consumed.
  On the third visit, a grass-fed beef burger (250 grams) will be consumed.
  Interventions: Dietary Supplement: Grain-Fed Beef Hamburger; Dietary Supplement: Grass-Fed Beef Hamburger; Dietary Supplement: Impossible BurgerTM
- Sequence 5: Grain-Fed, Impossible, Grass-Fed (Active Comparator): On the first visit, a grain-fed beef burger (250 grams) will be consumed.
  On the second visit, an Impossible BurgerTM (250 grams) will be consumed.
  On the third visit, a grass-fed beef burger (250 grams) will be consumed.
  Interventions: Dietary Supplement: Grain-Fed Beef Hamburger; Dietary Supplement: Grass-Fed Beef Hamburger; Dietary Supplement: Impossible BurgerTM
- Sequence 6: Grass-Fed, Impossible, Grain-Fed (Active Comparator): On the first visit, a grass-fed beef burger (250 grams) will be consumed.
  On the second visit, an Impossible BurgerTM (250 grams) will be consumed.
  On the third visit, a grain-fed beef burger (250 grams) will be consumed.
  Interventions: Dietary Supplement: Grain-Fed Beef Hamburger; Dietary Supplement: Grass-Fed Beef Hamburger; Dietary Supplement: Impossible BurgerTM

INTERVENTIONS:
Dietary Supplement: Grain-Fed Beef Hamburger — Bowl of grain-fed beef hamburger cooked without seasonings. 250 grams of uncooked hamburger weighed out, then cooked in a non-stick pan for 8 minutes, no seasoning or oils were used and rendered fat was poured into serving bowl.
Dietary Supplement: Grass-Fed Beef Hamburger — Bowl of grass-fed, grass-finished beef hamburger cooked without seasonings. 250 grams of uncooked hamburger weighed out, then cooked in a non-stick pan for 8 minutes, no seasoning or oils were used and rendered fat was poured into serving bowl.
Dietary Supplement: Impossible BurgerTM — Bowl of plant-based Impossible burger cooked without seasonings. 250 grams of uncooked Impossible burger weighed out, then cooked in a non-stick pan for 8 minutes, no seasoning or oils were used and rendered fat was poured into serving bowl.

SUMMARY:
The purpose of this study is to determine the effects of meat on inflammatory and metabolite profiles in middle-aged individuals after an acute meal. Up to 36 adults, who are overweight or obese and between 30-60 years old will undergo a consent/screening visit, followed by three study visits. On separate visits to the clinical research facilities at the Center for Human Nutrition Studies, participants will consume either 9 oz (250 grams) of cooked grain-fed beef, grass-fed beef, or a plant-based meat alternative (Impossible Burger). Blood will be drawn prior to food consumption and three more times after eating the meal at 1h, 3h, and 5h after participants finishing their meal. The investigators will use those blood samples to determine the impacts of these foods on inflammatory markers and metabolite profiles (compounds that circulate in our blood such as amino acids, fatty acids, and phenolics).

DETAILED DESCRIPTION:
BACKGROUND

An increasing number of people is interested in consuming either grass-fed beef or plant-based beef alternatives, such as the Impossible BurgerTM or Beyond MeatTM, believing that these choices are beneficial for consumer health; however, little to no work has been performed to study these beliefs and claims. The purpose of this study is to evaluate effects of plant-based meat, grass-fed beef, and grain-fed beef on postprandial plasma inflammatory and metabolite profiles in middle aged adults (30-60 y old). This work will offer new insight into manipulating the acute, post-meal inflammatory state by consumer food choices. It will also provide more insight how food-derived metabolites impact systemic metabolites in the human body through metabolomics analysis. This study will utilize a randomized cross-over design and every participant will consume each type of meat on three separate occasions separated by a minimum of three days.

STUDY OBJECTIVES

* To determine the effects of consuming 9 oz of the Impossible BurgerTM, grass-fed beef, or grain-fed beef on 300 min postprandial plasma inflammatory markers (IL-6, TNF-α, C-reactive protein, and VCAM-1).
* To determine effects on plasma metabolites (vitamin and mineral derivatives, polyphenols, amino acids etc.) collected through regular blood sampling during the 300 min postprandial phase (at 60 min, 180 min, and 300 min).
* To determine the effects on subjective satiety at 15, 30, 60 min and every hour thereafter following consumption.

DESIGN AND PROCEDURES

Participants will be asked to complete one screening/consent visit and three testing visits throughout their participation in the study. All visits will take place in clinical research space located at the Center for Human Nutrition Studies (CHNS) at Utah State University.

Phone Screen (Week 1. Duration: 15 min): Interested participants will be pre-screened by telephone, using a scripted list of questions (see attached) to identify individuals that may be eligible for study entry. Suitable candidates will then be provided a REDCap survey link to complete additional screening questions that asks them further details about their health, dietary habits, and sleep habits (see inclusion/exclusion criteria). Only the minimum PHI will be collected to determine eligibility. Responses will be reviewed by a study team member (all study team members will have completed the necessary CITI training) and potentially eligible candidates will be contacted to schedule a consent/screening visit. The pre-screen is put in place to confirm that the participant meets most of the inclusion/exclusion criteria before the subject is scheduled for a consent meeting. The phone screen is thus performed to limit the amount of ineligible research participants that are consented/screened that could easily be excluded by means of a phone screening. This would also provide interested participants with the opportunity to ask additional questions about the study and to determine if they are interested in moving forward with a consent/screening visit. This will limit both subject and research staff time burden.

Consent Visit (Week 1. Duration: 1 hour): This visit can be done virtually through Zoom or occur in person in the Center for Human Nutrition Studies (CHNS) at Utah State University. Potential subjects will attend a consent session conducted by a trained member of the research staff to present the details of the study. Interested participants will complete the informed consent process privately with study staff. The investigators will allow up to 60 minutes for the subjects to read the consent and ask questions. If a subject wants additional time to think about the study, this will be allowed. The study team will contact the subject three days after the initial consent visit ask if he or she has come to a decision. No study procedures will take place before written consent is obtained. To minimize subject burden, participants will be instructed during the phone screen that they have to opportunity to combine the consent visit with their screening visit (see below). If participants wish to combine visits, they are instructed that they will have to perform this visit in the morning after an overnight, 12-hour fast.

Screening Visit (Week 1. Duration: 1 hour): This visit will take place at the Center for Human Nutrition Studies (CHNS) and will last approximately 1 hour. The investigators ask participants to come in during the morning after an overnight, 12-hour fast. During this visit the following procedures will be performed:

* Blood Draw: A trained phlebotomist (the PI) will draw a fasted blood sample for routine blood work (see table 2 below) to ensure the participant qualifies for the study. Using a small needle, 12 ml blood will be collected from a vein in the participant's forearm or hand. Blood samples will be sent to LabCorp to be analyzed for HbA1C, Glucose, Basic Metabolic Panel (BMP), and Lipid panel. The blood of women of childbearing potential will be subject to a pregnancy test (hCG) as part of this screening blood draw. This will also occur through LabCorp.
* Body mass and height. Height (cm) will be measured without shoes. Body mass (kg) will be measured without shoes, coats, or sweaters. BMI will be calculated as body mass (kg) / height (m)2.
* Blood pressure: A blood pressure measurement will be taken using an automated upper arm blood pressure monitor (Omron BP5250). A total of three measurements will be taken and the average value of those will be collected for participant characterization.
* Questionnaires: Participant will be given a three-day food and sleep log to fill out for three days prior to each of the metabolic visits described below. The participant will also be given a food frequency questionnaire once at the beginning of the study, which will ask them about how often they consume animal products and if they are any of the following: "grass-fed, organic, pasture-raised, or bought on a farmers market". This will give us an indication of the habitual consumption of pasture-raised animal products of the participants. The food frequency questionnaire that will be used is a modified version of the Diet History Questionnaire III (NIH) with a 5-point ordinal scale as adapted from Baudry et al. (2015) (see attachment). The questionnaire reviews food and beverages typically consumed over the past year and takes approximately 30 minutes to complete.

Metabolic visits (Weeks 2-4. Number of Visits: 3. Duration: 7 hours each): These three visits will take approximately 7-hours each and will take place at The Center for Human Nutrition Studies (CHNS). Visits will be at least 3 days apart. Participants are required to fast for 12 hours prior to reporting to the laboratory. During this, participants will complete the following:

* Meat consumption: Using a randomized cross-over design, participants will ingest 250 g (9 oz) of an Impossible BurgerTM burger (plant), a grain-fed beef burger (grain-fed), a grass-fed beef burger (grass-fed). The meat will be stored as 9 oz. (250 g) patties in designated food freezers (-40 °C) in the NDFS kitchen and thawed overnight in a refrigerator (4 °C) prior to the subject's arrival the next morning. The meat will be cooked on a griddle in the CHNS metabolic kitchen on each side until an instant-read meat thermometer registers an internal temperature of 160 °F (71 °C). The patties will then be immediately served to the participant. Participants are provided with a standardized amount of water (1.5 liters) to drink during the 300 min post-meal phase. Participants will be asked to eat and drink the water at a comfortable rate but to try and finish within 30 min. No other food is allowed to be consumed during the ensuing 300 min postprandial phase. No other liquids are allowed to be consumed during that time as this would interfere with our protocol (see urine collection below). Subjects are also expected to remain seated in a chair during this time and can work/read/or watch entertainment on their own electronic device. Participants will be allowed to get up and use the rest-room; however, the investigators will ask participants to remain sedentary otherwise.
* Blood Draws: An intravenous catheter (IV) will be temporarily placed into a forearm or hand vein by a trained member of the study team (the PI) to collect repeated blood samples. The catheter will remain viable by a slow drip of saline. The investigators will collect four samples total (10 mL each; 40 mL or 2 ½ tablespoons) on each of the three metabolic visits. One sample will be collected right before participants eat and three more samples will be collected at 60, 180 min and 300 min after they consume the meal. These draws will be taken in a private room in clinical facilities, in a reclining leather chair. Participants will be provided with their clinical lab results that will be obtained from LabCorp. Results from bloodwork will be shared with participants via encrypted email using a USU email account.
* Urine Collection: A baseline urine sample will be collected prior to food consumption. Participants are asked to completely empty their bladder prior to food consumption. After food consumption, all urine will be collected in a urine jug (a 3000 mL urine collection bottle) during the 300-minute postprandial phase to study metabolites in the urine. All urine collections will be done by the participant themselves in private restroom facilities.
* Satiety Scale: Participants are asked to mark a validated satiety scale at 30, 60, 90, 120 min, and every hour thereafter until 300 min to assess subjective satiety after meat consumption.

Dietary and activity control: The investigators will ask participants to maintain their habitual diet, physical activity, and sleep levels.TThe investigators will ask participants to fill in 3-day dietary and sleep logs for the three days prior to their metabolic visit (see attachments). The investigators will also ask them to refrain from alcohol and strenuous physical activity (running, weightlifting etc.) for 2 days prior to each metabolic visit. The dietary and sleep logs will give the investigators insight if lifestyle factors leading up to each visit were similar and are likely to promote compliance to ensure robust biomarker results (inflammatory cytokines and metabolomics). Participants are asked to replicate their 3-day foods logs and sleep schedule as much as possible prior to each visit. Participants are also asked to not consume red meat or soy (main ingredient of plant burger) the day before each visit. This is done to minimize any prior presence of common red meat and soy-derived metabolites in the urine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥30 and ≤60 years;
* BMI ≥25 and ≤35 kg/m2;
* Weight stable in last 3 months (Loss or gain <4%);
* Hemoglobin A1C (HbA1C) ≤6.4%;
* Fasting plasma glucose concentration <126 mg/dl;
* Subjects must be able to speak and understand English to participate in this study

Exclusion Criteria:

* Use of medications that are known to affect the study outcome measures (e.g., NSAIDs, corticosteroids) or increase the risk of study procedures (e.g., anticoagulants) that cannot be temporarily discontinued for this study;
* Consuming >14 drinks per week;
* Use of cigarettes (or other tobacco products) in last 3 months;
* COVID vaccine within the last two weeks;
* Engaged in high-level competitive exercise (e.g., triathlon, marathon, powerlifting);
* Any inflammatory diseases(e.g. autoimmune diseases, coeliac disease, glomerulonephritis, hepatitis, inflammatory bowel disease, arthritis);
* Diagnoses of active malignancy, congestive heart failure, diabetes mellitus and/or chronic obstructive pulmonary disease;
* Use of antibiotics in last 60 days;
* Pregnant (or planning to in the next month) or lactating women;
* Soy allergy;
* Subjects who the study PI considers unable to safely complete the study protocol;
* Persons who are not able to grant voluntary informed consent;
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits;
* Vegetarian

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cytokine biomarker (IL-6) concentrations in plasma samples | Change from fasting concentrations after eating.
  Inflammatory biomarker concentrations of IL-6 (pg/ml) will be measured using ELISA kits at the Center for Human Nutrition Studies at Utah State University. Blood samples will be obtained via phlebotomy before the consumption of the meal, and at time points 60 minutes, 180 minutes, and 300 minutes after consumption of the meal, centrifuged immediately and stored at -80ºC until analyses are performed.
Inflammatory cytokine biomarker (C-reactive protein) concentrations in plasma samples | Change from fasting concentrations after eating.
  Inflammatory biomarker concentrations of C-reactive protein (CRP; ng/ml) will be measured using ELISA kits at the Center for Human Nutrition Studies at Utah State University. Blood samples will be obtained before the consumption of the meal, and at time points 60 minutes, 180 minutes, and 300 minutes after consumption of the meal, centrifuged immediately, and stored at -80ºC until analyses are performed.
Inflammatory cytokine biomarker (TNF-alpha) concentrations in plasma samples | Change from fasting concentrations after eating.
  Inflammatory biomarker concentrations of TNF-alpha (pg/ml) will be measured using ELISA kits at the Center for Human Nutrition Studies at Utah State University. Blood samples will be obtained before the consumption of the meal, and at time points 60 minutes, 180 minutes, and 300 minutes after consumption of the meal, centrifuged immediately, and stored at -80ºC until analyses are performed.
Inflammatory cytokine biomarker (Vascular Adhesion Molecule-1) concentrations in plasma samples | Change from fasting concentrations after eating.
  Inflammatory biomarker concentrations of Vascular Adhesion Molecule-1 (ng/ml) will be measured using ELISA kits at the Center for Human Nutrition Studies at Utah State University. Blood samples will be obtained before the consumption of the meal, and at time points 60 minutes, 180 minutes, and 300 minutes after consumption of the meal, centrifuged immediately, and stored at -80ºC until analyses are performed.
Relative abundance of metabolites in plasma samples using triple quad LC/MS-MS | Change from fasting concentrations after eating.
  Relative abundance (arbitrary units) of plasma metabolites after each meal will be measured using high-performance liquid chromatography tandem mass-spectrometry (LC/MS-MS). This analysis allows the simultaneous high-resolution measurement of a broad range of metabolites and will give insight into how food-derived metabolites from different meals impact metabolic pathways of human health. Blood samples will be obtained before each meal, and three times after the meal is consumed at time 60 minutes, 180 minutes, and 300 minutes, and centrifuged immediately and stored at -80ºC until analyses are performed. Multivariate statistical analysis and Partial least squares Discriminant Analysis will be used to identify features changed over time for each meal.

SECONDARY OUTCOMES:
Satiety Questionnaire | Immediately before meal
  Pre-Meal Satiety Question:
  Choose the best choice considering you have not yet eaten the test meal and you have arrived fasting, eating and drinking nothing but water since yesterday evening.
  Very Hungry; Hungry; A Little Hungry; No Particular Feeling; Somewhat Satisfied; Satisfied; Very Full.
Taste Questionnaire | Immediately after eating
  After finishing eating, answer the following questions.
  Q: 1. How strong is your desire to eat right now? A: 0-100 scale Not at all strong -- Extremely strong
  Q: 2. How pleasant is the taste of the meal? A: 0-100 scale Not at all pleasant -- Extremely pleasant
  Q: 3. How sweet does the meal taste? A: 0-100 scale Not at all sweet -- Extremely Sweet
  Q: 4. How salty is the taste of the meal? A: 0-100 scale Not at all salty -- Extremely salty
  Q: 5. How filling do you think the meal will be? A: 0-100 scale Not at all filling -- Extremely filling
  Q: 6. How familiar do you think the meal will be? A: 0-100 scale Not at all familiar -- Extremely familiar
  Q: 7. Overall, how did you feel about the flavor of the meal? A: 0-100 scale Disliked Extremely -- Liked Extremely
  Q: 8. How many calories do you think this meal has? A: 0-100 scale No calories at all -- Extremely high in Calories
Mood Questionnaires | Change in mood scores from baseline after eating.
  Mood Rating Survey
  Q: 1. How happy do you feel right now? A: 0-100 scale Not at all happy -- Extremely happy
  Q: 2. How much food could you eat right now? A: 0-100 scale Nothing at all -- The most I have ever eaten
  Q: 3. How full do you feel right now? A: 0-100 scale Not at all full -- Extremely full
  Q: 4. How hungry do you feel right now? A: 0-100 scale Not at all hungry -- Extremely hungry
  Q: 5. How thirsty do you feel right now? A: 0-100 scale Not at all thirsty -- Extremely thirsty
  Q: 6. How strong is your desire to eat right now? A: 0-100 scale Not at all strong -- Extremely strong
  Q: 7. How alert do you feel right now? A: 0-100 scale Not at all alert -- Extremely alert
  Q: 8. How clear-headed do you feel right now? A: 0-100 scale Not at all clear-headed -- Extremely clear-headed
  . These questions will be asked 30, 60, 90, 120, 180, 240, and 300 minutes after meal consumption

CONTACTS AND LOCATIONS:
Overall Officials: Stephan van Vliet, PhD, Principal Investigator — Utah State University
Locations (1):
- Center for Human Nutrition Studies, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol is attached to the ClinicalTrials.gov. Any collected data through RedCap and wet-lab assays will be made available upon publication. The metabolomics data will be deposited on Metabolomics Workbench (or a comparable repository) upon submission for publication.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Study protocol is available immediately. The analytical data will be available upon publication.
Access Criteria: Freely available.

REFERENCES:
- [Derived] Cloward J, Mason O, DeJesus I, Broadbent J, Payne T, Wengreen HJ, van Vliet S. Comparing postprandial inflammatory responses to a plant-based meat alternative, grass-finished beef, and grain-finished beef in healthy middle-aged adults: a 3-group randomized crossover trial. Am J Clin Nutr. 2026 Jan 8;123(3):101192. doi: 10.1016/j.ajcnut.2026.101192. Online ahead of print. PMID 41519303
- See also: Center for Human Nutrition Studies — https://caas.usu.edu/facilities/human-nutrition-studies

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT05690061/Prot_SAP_000.pdf